CLINICAL TRIAL: NCT01099163
Title: Effect of Conjugated Linoleic Acid Alone and in Conjunction With Vitamin E on Insulin Sensitivity, Beta Cell Function, Markers of Inflammation, Body Fat Mass and Other Biochemical Indicators in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Conjugated Linoleic Acid Alone and in Conjunction With Vitamin E in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Reza Rastmanesh, Ph.D, National Nutrition and Food Technology Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2387
Record Dates: First submitted 2010-04-05; First posted 2010-04-06 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes mellitus; CLA; Antioxidant; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 3g CLA (Experimental): 3 g CLA (50:50%) AND other diabetes medication currently prescribed to participant, 100 IU vitamin E
  Interventions: Dietary Supplement: Tonalin SG1000T FFA
- 3 g CLA (Active Comparator): 3 g CLA (50:50%) AND other diabetes medication currently prescribed to participant, vitamin E placebo
  Interventions: Dietary Supplement: Tonalin SG1000T FFA
- 3 g MCT + vit E placebo (No Intervention): 3 g MCT AND other diabetes medication currently prescribed to participant, 100 IU vitamin E placebo

INTERVENTIONS:
Dietary Supplement: Tonalin SG1000T FFA
  Arms: 3 g CLA; 3g CLA

SUMMARY:
Conjugated linoleic acids (CLAs) comprise a family of linoleic acid (18:2n-6; LA) isomers that are formed by biohydrogenation and oxidation processes in nature. The main form of CLA, cis-9, trans-11-18:2, can be produced directly by bacterial hydrogenation in the rumen or by delta-9 desaturation of the co-product vaccenic acid (trans-11-18:1) in most mammalian tissues including man. The second most abundant isomer of CLA is the trans-10, cis-12-18:2 form. Observations clearly emphasize that differences exist between mammalian species in their response to CLAs with mice being the most sensitive. The majority of studies on body compositional effects (i.e. fat loss, lean gain), on cancer and cardiovascular disease attenuation, on insulin sensitivity and diabetes and on immune function have been conducted with a variety of animal models. Recent studies indicate that some but not all of the effects observed in animals also pertain to human volunteers. Reports of detrimental effects of CLA intake appear to be largely in mice and due mainly to the trans-10, cis-12 isomer. Suggestions of possible deleterious effects in man due to an increase in oxidative lipid products (isoprostanes) with trans-10, cis-12 CLA ingestion require substantiation. Unresponsiveness to antioxidants of these non-enzymatic oxidation products casts some doubt on their physiological relevance. We hypothesized that supplementation with CLA + an antioxidant (vitamin E) in patients with diabetes mellitus may have beneficial effects on glycemic control and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus > 5 years
* HbA1c ≤ 9%
* Overweight or obese (BMI ≥ 25 kg/m2 and ≤ 30 kg/m2)
* Age ≥ 30 and ≤ 70 years (postmenopausal if female)
* Stable medical therapy for past 3 months
* Stable serum glucose for past 3 months (128-180 mg/Dl)
* Age between 30 to 50
* Use of metformin
* TG < 240 mg/Dl
* No alcohol, no insulin, no smoke
* No pregnancy, no menopause

Exclusion Criteria:

* Personal history of coronary heart disease
* Cerebrovascular disease or vascular disease
* Renal or hepatic disease
* Inflammatory diseases and thyroid diseases within the last years
* Use of drugs known to affect glycemic control, beta blockers, any change in daily activity profile, and diet

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2010-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity
beta cell function
glycosylated hemoglobin

SECONDARY OUTCOMES:
inflammatory mediators (TNF-alpha, Il-1beta, Il-6, CRP, adiponectin, leptin)
systolic and diastolic blood pressure
serum lipids (TG, LDL, HDL, LDL/HDL, ApoB100)
fibrinogen, PAI-1
body fat using bioimpedance
oxidative stress (MDA)

CONTACTS AND LOCATIONS:
Locations (1):
- Taleghani Hospital, Tehran, Tehran Province, Iran